CLINICAL TRIAL: NCT06003244
Title: Effect of Supplemental Oxygen Therapy (SOT) in Patients With Pulmonary Vascular Diseases (PVD) Defined as Pulmonary Arterial Hypertension or Chronic Thromboembolic Pulmonary Hypertension (PH) Who Permanently Live >2500m on 6-minute Walk Distance (6MWD)
Brief Title: High Altitude (HA) Residents With Pulmonary Vascular Diseases (PVD), 6 Minute Walk Distance (6MWD) Assessed at 2840m (HA) With and Without Supplemental Oxygen Therapy (SOT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PVD_HA_SOT_6MWD
Record Dates: First submitted 2023-08-10; First posted 2023-08-21 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Pulmonary Vascular Disease; Pulmonary Artery Hypertension; Chronic Thromboembolic Pulmonary Hypertension
Keywords: Pulmonary Hypertension; Hypoxia; Supplemental Oxygen Therapy; Pulmonary arterial hypertension; Chronic Thromboembolic Pulmonary Hypertension; High altitude; Pulmonary vascular disease
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension; Hypertension, Pulmonary; Hypoxia; Pulmonary Arterial Hypertension; Altitude Sickness

STUDY DESIGN:
Intervention Model Description: Each participant works as its own perfect control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ambient air (Active Comparator): Patient will perform tests on ambient air at 2840 m
  Interventions: Other: 6-minute walk distance (6MWD) test
- SOT via nasal canula (Experimental): Supplemental oxygen therapy (SOT) at 3l/min will be provided via a nasal cannula from a small oxygen bottle carried on the back according to standard care
  Interventions: Other: 6-minute walk distance (6MWD) test with supplemental oxygen (3 l/min, nasal)

INTERVENTIONS:
Other: 6-minute walk distance (6MWD) test — 6-minute walk distance (6MWD) test will be performed according to clinical standards
  Arms: Ambient air
Other: 6-minute walk distance (6MWD) test with supplemental oxygen (3 l/min, nasal) — 6-minute walk distance (6MWD) test will be performed according to clinical standards additionally with supplemental oxygen therapy (3l/min, nasal)
  Arms: SOT via nasal canula

SUMMARY:
The investigators aim to study the effect of SOT in participants with pulmonary vascular diseases (PVD) defined as pulmonary arterial hypertension or chronic thromboembolic pulmonary hypertension (PH) who permanently live >2500m on 6-minute walk distance (6MWD) assessed at 2840m.

DETAILED DESCRIPTION:
Participants with PVD diagnosed with precapillary PH with right heart catheterization and classified to groups 1 and 4 (PAH or CTEPH) who permanently live at HA >2500 (PVDHA) will have 6-minute walk distance near their living altitude in Quito at 2840m with and without SOT at 3l/min via nasal cannula according to a randomized cross-over design.

ELIGIBILITY:
IInclusion Criteria:

* Adult patients 18-80 years old of both genders,
* Residence > 2500m of altitude
* diagnosed with precapillary PH (mean pulmonary artery pressure (mPAP) >20 mmHg, pulmonary artery wedge pressure (PAWP) ≤15 mmHg and pulmonary vascular resistance (PVR) ≥2 wood units (WU) by right heart catheterization) with PH being classified as PAH or CTEPH according to guidelines
* Patients stable on therapy
* New York Heart Association (NYHA) functional class I-III
* Provided written informed consent to participate in the study.

Exclusion Criteria:

* Age <18 years or >80 years
* unstable condition
* Patients who cannot follow the study investigations, patient permanently living < 2500m.
* Patients with moderate to severe concomitant lung disease (FEV1<70% or forced vital capacity <70%), severe parenchymal lung disease, severe smokers (>20 cigarettes/day)
* Severely hypoxemic patients at Quito permanently have persistent oxygen saturation by pulseoximetry (SpO2) <80% on ambient air.
* Patients with chronic mountain sickness (Hemoglobin > 19 g/dl in women, >21 g/dl in men)
* Patient with a non-corrected ventricular septum defect
* Relevant concomitant other disease of the heart, kidney, liver, blood (anemia hemoglobin<11 g/dl)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-09-23 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
6-minute walk distance (6MWD) with supplemental oxygen therapy (SOT) vs. ambient air at 2840m | after 6 minute
  Change in 6MWD in meter between SOT 3l/min via nasal cannula vs. ambient air at 2840m

SECONDARY OUTCOMES:
SpO2 at rest and peak 6MWD with SOT vs. ambient air at 2840m | 6 minutes
  Change of the arterial oxygen saturation by pulseoximetry (SpO2) at rest and at peak 6MWD with SOT 3l /min vs. ambient air at 2840 m
Heart rate at rest and peak 6MWD with SOT vs. ambient air at 2840m | 6 minutes
  Change of heart rate (bpm) at rest and at peak 6MWD with SOT 3l /min vs. ambient air at 2840 m
Blood pressure at rest and peak 6MWD with SOT vs. ambient air at 2840m | 6 minutes
  Change of Blood pressure (mmHg) at rest and at peak 6MWD with SOT 3l /min vs. ambient air at 2840 m
Borg dyspnea scale at rest and peak 6MWD with SOT vs. ambient air at 2840m | 6 minutes
  Change of Borg dyspnea scale at rest and at peak 6MWD with SOT 3l /min vs. ambient air at 2840 m

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Ulrich, Prof. Dr., Principal Investigator — University Hospital Zurich, Departement of Pulmonology; Rodrigo Hoyos, Dr., Principal Investigator — Carlos Adrade Marin Hospital of Quito, Equador
Locations (1):
- University Hospital Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Data will be provided upon request and based on a clear intention reviewed by an ethical review board.